CLINICAL TRIAL: NCT01270906
Title: A Phase 1 Dose Escalating Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodyniamics of CHIR-258 in Subjects With Advanced Solid Tumor Malignancies
Brief Title: Safety of CHIR-258 (TKI258) in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Chiron Corporation (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2101 (CHIR-258-001)
Record Dates: First submitted 2010-12-02; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Neoplasms; Cancer; Tumors
Keywords: Neoplasms; Cancer; Tumors; Administration; oral; CHIR258; CHIR-258; CHIR 258; TKI258; TKI-258; TKI 258; dose finding
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- CHIR-258 (TKI258) (Experimental)
  Interventions: Drug: CHIR-258 (TKI258)

INTERVENTIONS:
Drug: CHIR-258 (TKI258)

SUMMARY:
Phase I dose finding study in solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically documented, advanced-stage, primary or metastatic solid tumors that are refractory to standard therapy or for which no curative standard therapy exists.
* Evidence of measurable or evaluable disease.
* All acute toxic affects of any prior radiotherapy, chemotherapy, or surgical procedures must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 3.0) Grade ≤1; surgery must have occurred at least 28 days prior to study enrollement.
* Age must be at least 18 years.
* Last dose of antineoplastic therapy (except for hormonal therapy) must be more than 21 days; subjects may continue to receive luteinizing hormone-releasing hormone analog therapy for prostate cancer.
* ECOG performance status must be 0 or 1.
* Life expectancy of at least 3 months.
* Patient must meet protocol-specified laboratory values.

Exclusion Criteria:

* Concurrent therapy with any other investigational agent.
* Intracranial edema, intracranial metastasis, or epidural disease.
* Pregnant or breastfeeing women. Female subjects must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male subjects must agree to use effective contraception or be surgically sterile. The definition of effective contraception will be based on the judgment of the investigator or a designated associate. All at-risk female subjects must have a netative pregnancy test (serum or urine) within 10 days prior to the start of study treatment.
* Clinically significant cardiac disease (New York Heart Association Class III or IV) including pre-existing arrhythmia, congestive heart failure, cardiomyopathy, or subjects with baseline mean QTc interval greater than 450 msec (males) and 470 msec (females) or grade 2 or higher compromised left ventricular ejection fraction (LVEF) as determined by MUGA or ECHO.
* Dementia or altered mental status that would prohibit informed consent.
* Diabetes mellitus (insulin-dependent or -independent disease requiring chronic medication).
* Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring two or more interventions/month.
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities (nausea, diarrhea, vomitting) with toxicity greater than NCI CTCAE grade 2.
* Prior acute or chonic pancreatitis of any etiology.
* Prior intra-or extra-hepatic biliary obstruction wtihin the previous 12 months or history of malignant obstruction requiring a bilary stent, unless stably treated with no prior obstruction or blockage of the stent.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study-drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, make the subject inappropriate for this study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
dose limiting toxicity (DLT) to define the maximum tolerated dose (MTD). The DLT is defined as treatment related grade 3 or grade 4 adverse events or abnormal lab test that occurred in the first 28 days after start of study drug. | continuous monitoring for the first 28 days after start of the study medication

SECONDARY OUTCOMES:
characterize pharmacokinetic (PK) profile of study drug after single and repeated doses. The PK profile includes maximum blood concentration (Cmax) and time to reach maximum blood concentration (Tmax). | day 1 and day 15 at the following timepoints: pre-drug and 30 minutes, 1, 2, 3, 4, 5, 6, and 8 hours after dose
Pharmacodynamics (PD) in terms of serine-threonine kinase phosphorylation inhibition in blood before and after dose | day 1 and day 15 at the following timepoints: pre-drug, 4 and 24 hours after dose
Antitumor activity by comparing baseline and post-treatment changes. Tumor assessment will be performed using the Response Evaluation Criteria in Solid Tumors (RECIST) | baseline and once every two months thereafter
urinary metabolic profiling - examination of the ratio of beta-hydroxycortisol/cortisol | 24 hour urine collection on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Sutton

REFERENCES:
- [Derived] Wang X, Kay A, Anak O, Angevin E, Escudier B, Zhou W, Feng Y, Dugan M, Schran H. Population pharmacokinetic/pharmacodynamic modeling to assist dosing schedule selection for dovitinib. J Clin Pharmacol. 2013 Jan;53(1):14-20. doi: 10.1177/0091270011433330. Epub 2013 Jan 24. PMID 23400739